CLINICAL TRIAL: NCT06088459
Title: Phase I Safety and Immunogenicity Study of NWRD06 in Hepatocellular Carcinoma Patients After Radical Resection
Brief Title: NWRD06 DNA Plasmid for HCC After Radical Resection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newish Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEWISH-GPC3-101
Record Dates: First submitted 2023-09-27; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Naked DNA Vaccine; GPC3
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: This study is divided into three dose groups climbed from low-dose group to high-dose group in turn according to the 3+3 dose escalation principle.
  Three dose groups were preset in this study: dose group 1 and low-dose group [a single dose of 1mg was administered three times at week 0, 4 and 8, respectively, with cumulative administration of 3mg]; Dose group 2, middle-dose group [single dose of 4mg, administered 3 times at week 0, 4, 8, respectively, cumulative administration of 12mg]; Dose group 3, high-dose group [a single dose of 8mg, administered at week 0, 4 and 8, a total of 3 times, cumulative administration of 24mg].
  After the completion of treatment, the subjects shall continue to receive safety follow-up until 28 days after the last administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NWRD06 by electroporation (Experimental): Patients will be assigned to three dose groups:1mg, 4mg, and 8mg. Each patient will be administered NWRD06 by electroporation in entire study period. The Maximum Tolerated Dose of NWRD06 will be determined by the classical 3+3 dose escalation schedule. The number of patients will be ranged from 9 to 18.
  Interventions: Biological: 1mg NWRD06 administered by electroporation; Biological: 4mg NWRD06 administered by electroporation; Biological: 8mg NWRD06 administered by electroporation

INTERVENTIONS:
Biological: 1mg NWRD06 administered by electroporation — DNA plasmid delivered via IM injection + electroporation using TERESA device
Biological: 4mg NWRD06 administered by electroporation — DNA plasmid delivered via IM injection + electroporation using TERESA device
Biological: 8mg NWRD06 administered by electroporation — DNA plasmid delivered via IM injection + electroporation using TERESA device

SUMMARY:
This is a dose escalation Phase 1 clinical study to evaluate the safety and immunogenicity of Glypican3 (GPC3)-targeted DNA plasmid vaccine (NWRD06) in patients with GPC3-positive primary hepatocellular carcinoma after radical resection.

DETAILED DESCRIPTION:
This study is divided into three dose groups:1mg, 4mg, and 8mg. Each patient will be administered NWRD06 by electroporation in entire study period. The Maximum tolerated dose of NWRD06 will be determined by the classical 3+3 dose escalation schedule. The number of patients will be ranged from 9 to 18.

After the completion of treatment, the subjects shall continue to receive safety follow-up until 28 days after the last administration.

Immunologic reactogenicity in blood samples was assessed at week 0, week 2, week 4, week 6, week 8, week 10, week 12.

Peripheral blood samples were then collected every 3 months for immunogenicity assessment until disease progression or specific immune response became undetectable or the study was withdrawn for various reasons or ended (whichever occurred first).

ELIGIBILITY:
Inclusion Criteria:

Patients had to meet all of the following inclusion criteria:

1. 18≤ age ≤60, regardless of gender;
2. Diagnosis of primary hepatocellular carcinoma (HCC) by pathohistological examination;
3. Immunohistochemical staining that was positive for GPC3;
4. Barcelona clinic liver cancer (BCLC) stage A/B or Chinese Hepatocellular carcinoma Stage (CNLC) Ib-IIIa;
5. Underwent radical resection of liver cancer (surgery, ablation) followed by hepatic artery interventional therapy before the first NWRD06 administration; The interval between radical resection and the first NWRD06 administration was less than 12 weeks, and the interval between hepatic artery interventional therapy and the first NWRD06 administration was more than 7 days;
6. No residual intrahepatic tumor was found by imaging examination within 4 weeks before the first NWRD06 administration; No lymph node metastasis, no extrahepatic metastasis;
7. Patients undergoing radical resection of liver cancer should meet the intraoperative criteria of radical resection of liver cancer:1)There was no invasion of adjacent organs, hilar lymph nodes or distant metastasis during the operation; 2) Negative cutting margin;
8. No Vp4 macrovascular invasion, hepatic vein or inferior vena cava macrovascular invasion of any grade after radical resection; Notes: Patients with VP1, VP2 and VP3 macrovascular invasion diagnosed via histopathologic examination or imaging test meet the inclusion criteria.
9. Within 1 week before the first NWRD06 administration, ECOG performance status score was 0-1;
10. Child-Pugh score A/B (≤7) within 1 week before the first NWRD06 administration;
11. Major organ functions were normal within 1 week before the first NWRD06 administration: 1) Blood routine: Hemoglobin (Hb) ≥90 g/L; Platelet count (PLT) ≥75×109/L; 2) The liver: Total bilirubin (TB) ≤3× upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5×ULN; Plasma albumin ≥30g/L; 3)Kidney: Serum creatinine (Scr) ≤1.5×ULN, or creatinine clearance ≥40 mL/min (serum creatinine > 1.5 x ULN);
12. The expected survival time is more than 6 months;
13. Patients with non-viral primary HCC meet the inclusion criteria. For patients with Hepatitis B virus-related primary HCC(HBV-HCC) or Hepatitis C virus-related primary HCC(HCV-HCC), antiviral therapies should be carried out simultaneously;
14. Within 1 week before the first NWRD06 administration, women of childbearing age must have a negative serum pregnancy test and consent to use effective contraception during the use of the study drug and within 6 months after the last administration of the study drug. For men, they should be surgically sterilized or agree to use effective contraception during study drug use and for 6 months after the last administration of study drug.
15. Have fully understood the study and voluntarily signed the ICF, have good communication with the investigator, and are able to complete all treatments, examinations, and visits stipulated in the study protocol.

Exclusion Criteria:

Patients with any of the following were excluded from the study:

1. HCC recurred or metastasis before the first NWRD06 administration;
2. Before the first NWRD06 administration, the investigator judged that the patient had not fully recovered from the toxicity and/or complications of radical resection;
3. Accompanied by hepatic encephalopathy;
4. Regular renal dialysis is required;
5. with uncontrolled pleural effusion, pericardial effusion, or moderate or more ascites (refers to ascites that cannot be easily controlled by diuretic treatment);
6. A history of gastrointestinal bleeding, current active bleeding, or bleeding tendency within 28 days before screening;
7. Had received systemic antitumor therapy (including chemotherapy, molecular targeted therapy, biological immunotherapy) for liver cancer within 28 days before screening;
8. Participated in another clinical trial or was under observation in another clinical trial within 28 days prior to screening;
9. Continuous (more than 1 week) glucocorticoid therapy (dose equivalent to prednisone > 10 mg/ day), except hormone replacement therapy and intratracheal administration;
10. A history of immune deficiency or autoimmune diseases (e.g., rheumatoid joint disease, systemic lupus erythematosus, multiple sclerosis, etc.);
11. A history of allogeneic stem cell/tissue/solid organ transplantation (including bone marrow transplantation);
12. With uncontrolled severe infection (> grade 2 NCI-CTCAE adverse events, version 5.0);
13. Patients with a history of human immunodeficiency virus (HIV) infection or carriers of syphilis;
14. Patients with serious other organ dysfunction or cardiopulmonary diseases;
15. Epilepsy that requires treatment with medication (e.g. steroids or antiepileptic drugs);
16. Had or currently has other malignancies (with the exception of adequately treated and completely cured ductal carcinoma in situ of the breast, carcinoma in situ of the cervix, basal cell carcinoma of the skin, superficial bladder tumor, or any malignancy that was cured more than 5 years before study entry);
17. A known history of albumin allergy, or severe allergy, or allergic disease, or allergic constitution, or severe iodine contrast allergy, meeting any of these criteria;
18. Severe mental illness;
19. A history of drug or alcohol abuse;
20. Pregnant or lactating women, or women of childbearing age with positive blood pregnancy tests;
21. Patients deemed by the investigator to be ineligible for this clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | From first administration of NWRD06 to 28 days after the last administration
  It would be determined based on the rate and severity grade of events or abnormalities through evaluating systemic or local adverse events, clinical laboratory test results, vital signs that is definitely, probably, or possibly related to the test drug occurring within 28 days of the last dosing will be classified as DLT during dosing climb.
All adverse events (AE) | 12 weeks
  All adverse events (AE) will be determined based on the rate and severity grade of events, including incidence and severity of serious adverse events (SAE) (according to NCI-CTCAE Standard version 5.0 of common Terms for Adverse Events)

SECONDARY OUTCOMES:
Immunogenicity | At week 0, week 2, week 4, week 6, week 8, week 10, week 12 and then collected every 12 weeks until disease progression or specific immune response became undetectable or the study was withdrawn for various reasons or ended (whichever occurred first).
  GPC3 specific immune response in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Hong, Ph.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication
Access Criteria: by publication